CLINICAL TRIAL: NCT02116985
Title: Dual-Loop Target Controlled Infusion of Propofol and Remifentanil Guided by Narcotrend Index in Laparoscopic Cholecystectomy
Brief Title: Dual-Loop Target Controlled Infusion in Laparoscopic Cholecystectomy (DLTCI)
Acronym: DLTCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: dual-loop
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Cholecystolithiasis
Keywords: Dual-Loop TCI; NI; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual-Loop TCI (Experimental): the controller in the current study measures and calculates the error(NI error),which is the difference between the set point(NI=36)and the measured NI.If the NI error is different from 0,the controller determines a new propoflo and/or remifentanil concentration.
  Interventions: Device: Dual-loop TCI
- manual (Placebo Comparator): the investigator modified the effect-site target concentrations of both drugs without minimum or maximum concentration limits without using the Narcotrend monitor only depend on the experience of anesthesiologist.
  Interventions: Device: manual

INTERVENTIONS:
Device: Dual-loop TCI — the controller in the current study measures and calculates the error(NI error),which is the difference between the set point(NI=36)and the measured NI.If the NI error is different from 0,the controller determines a new propoflo and/or remifentanil concentration.
  Arms: Dual-Loop TCI
Device: manual — the investigator modified the effect-site target concentrations of both drugs without minimum or maximum concentration limits without using the Narcotrend monitor only depend on the experience of anesthesiologist.
  Arms: manual

SUMMARY:
Laparoscopic Cholecystectomy applied to Artificial pneumoperitoneum and the extent of Surgical stimulation cause the wave of hemodynamics increase vigorously, which make it difficult to judge the depth of anesthesia according to traditional hemodynamics index such as heart rate and blood pressure.In case of this, the investigators design this research to study the Closed-Loop Target Controlled Infusion to anaesthesia of individualization guided by a Narcotrend index monitor in Laparoscopic Cholecystectomy.

DETAILED DESCRIPTION:
Anesthetics alter electrocortical activity in a dose-dependent manner,and it is suggested that electroencephalographic(EEG)activity can provide a reliable basis for a surrogate measurement of hypnosis.An EEG monitor,the Narcotrend Index(NI),has proven useful to titrate hypnotic drugs.Because it is a single composite measure monitored continuously,it has been used in controlled studies to automatically guide propofol administration.Conversely,automated delivery systems for opioids have seldom been described using EEG activity There are no specific measures to quantify analgesia directly.Nevertheless,in the interaction between opioid-hypnotic synergy and loss of consciousness,when the dose of analgesic administered is sufficient to inhibit autonomic response to noxious stimuli,then the required hypnotic concentration is only that needed to achieve loss of consciousness.Moreover,a noxious stimulus such as laryngoscopy or periosteal pressure to the tibia may cause electrocortical activation with an increase in Narcotrend index,which indirectly reflects the analgesic state or the level of antinociception.Finally,an excitatory EEG arousal reaction resulting from nociceptive stimulation can provide a rational basis for analgesia administration.It can then be hypothesized that Narcotrend index could also be the controlled variable for opioid administration.

ELIGIBILITY:
Inclusion Criteria:

1. require general anesthesia
2. expected to last>30 minutes
3. 18~90 years
4. ASA Ⅰ~Ⅳ level

Exclusion Criteria:

1. psychiatric illness
2. supraspinal neurological disorders
3. cranial neurosurgical procedures
4. patients equipped with a pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The total dose of propofol and remifentanil | within two hours from the beginning to the end of the propofol and remifentanil
  record the total dose of propofol and remifentanil from the beginning to the end of anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500